CLINICAL TRIAL: NCT07146984
Title: Application of PDCA Cycle in Tracheal Intubation Training for Emergency Medicine Residents
Acronym: PACT
Status: Enrolling by invitation | Type: Observational
Sponsor: Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Mai Xiaowei, Associate Chief Physician, Guangzhou Panyu Central Hospital
Other Study IDs: PYRC-2024-280-01
Record Dates: First submitted 2025-08-16; First posted 2025-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Tracheal Intubation; Medical Education
Keywords: PDCA cycle; emergency medicine; tracheal intubation; medical education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PDCA Cycle-Based Training Intervention: The Plan-Do-Check-Act (PDCA) cycle Based Training Intervention
  Interventions: Behavioral: Behavioral (Educational Training Program)

INTERVENTIONS:
Behavioral: Behavioral (Educational Training Program) — A structured training program for emergency medicine residents based on the Plan-Do-Check-Act (PDCA) cycle. The intervention includes didactic teaching, simulation-based airway management practice, supervised clinical intubation, iterative performance assessment, and feedback-driven improvement.

SUMMARY:
Tracheal intubation is a critical but technically demanding procedure in emergency airway management. Junior emergency medicine residents often struggle to achieve proficiency, leading to increased risks of complications. This study evaluates the effectiveness of a Plan-Do-Check-Act (PDCA) cycle-based training program in improving intubation skills.

The study was conducted in the emergency department of a tertiary teaching hospital. Residents performing intubations in 2023 with conventional training served as the control group, while those trained with the PDCA model in 2024 formed the intervention group. The PDCA program included structured lectures, high-fidelity simulation, supervised clinical practice, and iterative feedback.

Primary outcomes were first-attempt success rate and intubation completion time. Secondary outcomes included incidence of local airway trauma, extubation failure due to airway injury within 72 hours, and resident satisfaction. This study aims to provide evidence that PDCA-based training can enhance procedural competency, safety, and learner satisfaction in emergency airway management.

DETAILED DESCRIPTION:
Tracheal intubation is a high-risk, time-sensitive procedure that is fundamental to emergency airway management. Despite its lifesaving role, it remains one of the most technically challenging skills for junior emergency medicine residents. Failed or delayed intubation is associated with serious complications, including airway trauma, hypoxemia, aspiration, and cardiac arrest. Traditional didactic training often lacks the iterative practice and structured feedback required for durable skill acquisition.

The Plan-Do-Check-Act (PDCA) cycle is an educational quality improvement framework that emphasizes continuous evaluation, feedback, and refinement. This study was designed to investigate whether a PDCA-based training model could improve intubation competency among emergency medicine residents in a tertiary teaching hospital.

This prospective observational study compared intubation performance before and after PDCA cycle implementation. The control group included residents performing intubations in 2023 with conventional training, while the intervention group included residents trained with the PDCA model in 2024. The PDCA program consisted of structured didactic sessions, high-fidelity simulation, supervised clinical practice, and iterative debriefing with continuous feedback loops.

Primary outcomes were first-attempt success rate and intubation completion time, as these are widely recognized benchmarks of procedural safety and efficiency. Secondary outcomes included the incidence of local airway trauma, extubation failure due to airway injury within 72 hours, and resident satisfaction with training.

We hypothesized that PDCA-based training would significantly improve first-pass success, shorten intubation time, reduce airway-related complications, and enhance trainee satisfaction. The findings may provide evidence for adopting structured, feedback-oriented frameworks in emergency and critical care training, with broader implications for competency-based medical education.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine residents rotating in the emergency department during the study period.
* Residents who are required to perform tracheal intubation as part of clinical training.
* Residents who have completed baseline theoretical and simulation-based airway management training.
* Voluntary participation with written informed consent.

Exclusion Criteria:

* • Residents who refuse to participate or withdraw consent.

  * Residents with prior advanced airway fellowship training or extensive intubation experience (>50 independent intubations).
  * Residents who are unable to complete the full PDCA-based training program due to absence or rotation schedule.
  * Any medical condition or circumstance deemed by investigators to interfere with participation or data integrity.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Emergency medicine residents from the Department of Emergency, Panyu Central Hospital, Guangzhou Medical University, China. Participants were postgraduate residents rotating in the emergency department during the study period and were required to perform tracheal intubation as part of their clinical training.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
First-Attempt Success Rate of Tracheal Intubation | Within procedure (immediately at time of intubation)
  The proportion of tracheal intubation attempts by emergency medicine residents successfully completed on the first attempt, as verified by standard clinical confirmation (e.g., chest rise, end-tidal CO₂, auscultation, chest X-ray).

SECONDARY OUTCOMES:
Intubation Completion Time | Periprocedural (measured once during each intubation attempt, from laryngoscope insertion to confirmed tracheal tube placement, using a stopwatch
  Time in seconds from insertion of the laryngoscope to confirmation of successful tube placement.
Incidence of Local Airway Trauma | Assessment was performed immediately after completion of intubation and within 5 minutes post-procedure, by direct laryngoscopic visualization or suction catheter inspection
  Presence of fresh blood in the airway post-intubation, excluding bleeding from preexisting conditions (e.g, subglottic mass, pulmonary hemorrhage).
Extubation Failure Due to Airway Injury | Assessment was performed within 72 hours following planned extubation. Patients were monitored for the need of reintubation, and airway injury was confirmed by laryngoscopy when extubation failure occurred.
  Reintubation within 72 h despite meeting extubation criteria, confirmed by laryngoscopy (e.g., edema, vocal cord paralysis, granulation, or subglottic stenosis).
Mean Questionnaire Score on Learning Experience and Perceived Training Value | Immediately after completion of the training session (within 24 hours).
  Assessed via anonymous questionnaire administered immediately after training。Scores are reported on a 5-point Likert scale (1 = very poor, 5 = excellent), with higher scores indicating a better learning experience and greater perceived training value.

CONTACTS AND LOCATIONS:
Overall Officials: yingshen wen, Study Director — Department of emergency, The Affiliated Panyu Central Hospital, Guangzhou Medical University, China
Locations (1):
- The Affiliated Panyu Central Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT07146984/Prot_000.pdf
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT07146984/ICF_001.pdf